CLINICAL TRIAL: NCT06429748
Title: A Prospective Study to Evaluate Symptoms Following Repetitive Transcranial Magnetic Stimulation (rTMS)
Brief Title: Symptom Evaluation Following Repetitive Transcranial Magnetic Stimulation
Acronym: SET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 44-50019-000
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Neurologic Symptoms
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Open Label (Experimental): Single Group
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — repetitive Transcranial Magnetic Stimultion

SUMMARY:
A prospective study to evaluate symptoms following repetitive transcranial Magnetic stimulation.

DETAILED DESCRIPTION:
Open-label, multicenter, prospective pilot study conducted in an adult population receiving rTMS treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 22 to 70 years of age
2. Voluntarily provides written informed consent and agree to comply with study procedures, including attending all study visits and completing all study assessments.
3. Score > or = 8 on ISI scale
4. If subject is on any psychiatric or sleep medication, dose must be stable for two weeks prior to enrollment and remain stable throughout the trial.
5. If female, not breastfeeding, no known or suspected pregnancy, a status of nonchildbearing potential or use of an acceptable form of birth control.
6. Subject on stable dose regime for other concurrent medications like hormonal therapy for menopause transition etc.

Exclusion Criteria:

1. Subject meets any one or more of the contraindications for TMS Therapy per current treatment guidelines as determined by the PI.
2. History of head trauma associated with loss of consciousness or diagnosed as concussion.
3. History of fainting, syncope, hearing problems or ringing in the ears (tinnitus)
4. Has any metallic implant(s) in or near the head (e.g., pacemaker, defibrillator, neurostimulator, etc.) including any splinters, fragments, clips, etc.
5. Has an implanted stimulator device (including device leads) in or near the head. (e.g. deep brain stimulator, cochlear implant, vagus nerve stimulator.)
6. Has medication infusion device.
7. Subjects with any prior TMS or MRI complications, or any other issues/circumstance which, in the opinion of the investigator, might interfere with safety, study participation, or which might confound data interpretation.
8. PHQ-9 total score > or = 10 or QIDS total score > or = 11.
9. Drug abuse or dependence of the illicit substance. (Abuse or Dependence, as defined by DSM-V-TR)
10. Current diagnosis or known history of neurologic disease (e.g., epilepsy, convulsion, seizure)
11. Other known disorder (e.g., narcolepsy, a breathing-related sleep disorder like Obstructive Sleep Apnea, a circadian rhythm sleep-wake disorder, a parasomnia) as defined by DSM-V-TR.
12. Has a clinically significant abnormality on the screening examination.
13. Participation in any clinical trial with an investigational drug or device within the past month or concurrent with study participation.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in multiple symptoms after rTMS treatment. | 4 weeks
  Assess changes in multiple symptoms scores based on patient reported questionnaires from baseline to end of acute.

SECONDARY OUTCOMES:
Durability of changes in symptoms | 16 weeks
  Assess changes in multiple symptoms scores based on patient reported questionnaires from baseline to final follow-up visit.

OTHER OUTCOMES:
Safety Outcome | 16 weeks
  Treatment related Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Steve Erickson, Study Director — Neuronetics
Locations (1):
- Charlotte Skin and Laser, Charlotte, North Carolina, United States